CLINICAL TRIAL: NCT00176917
Title: Hematopoietic Stem Cell Transplantation for Hurler Syndrome, Maroteaux Lamy Syndrome (MPS VI), and Alpha Mannosidase Deficiency (Mannosidosis)
Brief Title: Stem Cell Transplantation for Hurler
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMN-MT1999-07; 0104M93821 (Other: IRB, University of Minnesota); NCT00005899 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Mannosidosis; Mucolipidosis Type II (I-cell Disease)
Keywords: stem cell transplant; storage disease; errors of metabolism
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis VI; Mannosidase Deficiency Diseases; Mucolipidoses | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Busulfan; Cyclophosphamide; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): All patients treated with chemotherapy and transplantation.
  Interventions: Procedure: Stem Cell Transplant; Drug: Busulfan, Cyclophosphamide, ATG

INTERVENTIONS:
Procedure: Stem Cell Transplant — The purpose of hematopoietic cell transplantation is to introduce hematopoietic cells from a normal donor that contains the enzyme able to get rid of the substances that have accumulated in the body of patients with storage diseases. Hematopoietic cells can come from bone marrow, peripheral blood (i.e., the blood circulating in our body's blood vessels) or umbilical cord blood (i.e. blood taken from the umbilical cord after a baby is born and umbilical cord is cut).
  Other Names: Bone Marrow Transplant
Drug: Busulfan, Cyclophosphamide, ATG — Prior to transplantation, subjects will receive BUSULFAN intravenously (IV) via the Hickman line twice daily for 4 days, CYCLOPHOSPHAMIDE intravenously via the Hickman line once a day for 4 days, and ANTI-THYMOCYTE GLOBULIN IV via the Hickman line twice daily for three days before the transplant. These three drugs are being given to help the new marrow "take" and grow. METHYLPREDNISOLONE will be given as a pre-medication for the ATG.
  Other Names: Busulfex, Cytoxan, Thymoglobulin

SUMMARY:
The purpose of this study is to determine the safety and engraftment of donor hematopoietic cells using this conditioning regimen in patients undergoing a hematopoietic (blood forming) cell transplant for Hurler syndrome, Maroteaux Lamy syndrome, Mannosidosis, or I-cell disease.

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive Busulfan intravenously (IV) via the Hickman line four times daily for 4 days, Cyclophosphamide intravenously via the Hickman line once a day for 4 days, and Anti-Thymocyte Globulin IV via the Hickman line twice daily for three days before the transplant. These three drugs are being given to subjects to help the new marrow "take" and grow.

On the day of transplantation, the donor's hematopoietic cells will be transfused via central venous catheter.

After hematopoietic cell transplant, subjects will then receive two drugs, cyclosporin and either methylprednisolone or Mycophenolate Mofetil (MMF). Cyclosporin and methylprednisolone or MMF are given to help prevent the complication of graft-versus-host disease and to decrease the chance that the new donor cells will be rejected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mucopolysaccharidosis, type I (e.g., Hurler syndrome), Maroteaux-Lamy syndrome (MPS VI), Alpha Mannosidosis, or mucolipidosis type II (I-cell disease) who have an HLA-identical or mismatched (at 1 antigen) related marrow, PBSC, or cord blood donor.
* Patients with Mucopolysaccharidosis, type I, Maroteaux-Lamy syndrome (MPS VI), Alpha Mannosidosis, or mucolipidosis type II (I-cell disease) who have an HLA-identical or HLA-1 antigen mismatched unrelated marrow, PBSC, or HLA-0-2 antigen mismatched umbilical cord blood donor.
* Patients with MPS type I, Maroteaux Lamy Syndrome (MPS VI), or mucolipidosis type II (I-cell disease) will have a mental developmental index within two standard deviations of the normal mean, as best as can be determined using Bayley scales of infant development or other standardized testing, recognizing that these may be affected by speech and/or hearing impairment.
* Adequate organ function:
* Cardiac: ejection fraction >40%; no decompensated congestive heart failure or uncontrolled arrhythmia
* Renal: serum creatinine <2.0 mg/dl
* Hepatic: total bilirubin <3x Upper limits of normal transaminases < 5.0 x Upper limits of normal
* Signed consent.

Exclusion Criteria:

* Presence of major organ dysfunction (see above)
* Pregnancy
* Evidence of HIV infection or known HIV positive serology
* Patients or parents are psychologically incapable of undergoing BMT with associated strict isolation or documented history of medical non-compliance
* Patients >50 kg may be at risk for having cell doses below the goal of ≥ 10 x 106 CD 34 cells/kg and therefore will not be eligible to receive unrelated PBSCs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-05; Primary Completion 2008-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transplant Patients: Patients that received hematopoietic stem cell transplant.
Period: Overall Study
Arm/Group | Transplant Patients
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Transplant Patients
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Donor Cells in Study Population (Chimerism).
Description: Donor-derived engraftment determined by restriction fragment length polymorphism (RFLP).
Time Frame: at 21 days, 42 days, 60 days, 100 days, 6 months, and 1 year
Population: Day 21 (24 patients included), Day 42 (15 pts), Day 60 (29 pts), Day 100 (25 pts), 6 Months (18 pts), 1 Year (16 pts).
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Transplant Patients
Number analyzed (Participants) | 41
Percentage
  21 Days Post Transplant | 85.8 (28.4)
  42 Days Post Transplant | 73.2 (31.6)
  60 Days Post Transplant | 84.6 (27.9)
  100 Days Post Transplant | 81.1 (26.8)
  6 Months Post Transplant | 81.6 (29.6)
  1 Year Post Transplant | 91.5 (18.8)

2. Secondary Outcome: Number of Patients Surviving on Study
Description: Number of patients surviving (alive) at specified timepoints.
Time Frame: at 100 days, 1 year, and 3 years post transplant
Population: Day 100 and 1 Year timepoints include all 41 patients. Year 3 includes 36 patients (5 pts not yet at followup timepoint.)
Measure: Number; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 41
Participants
  Day 100 Post Transplant | 37
  1 Year Post Transplant | 28
  3 Years Post Transplant | 27

3. Secondary Outcome: Number of Patients Who Failed Engraftment.
Description: Toxicity (undesireable effect) of hematologic donor cell engraftment is determined by failure to engraft at Day 42.
Time Frame: Day 42 Post Transplant
Population: 1 patient of 41 failed engraftment - per protocol.
Measure: Number; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 41
Participants | 1

4. Secondary Outcome: Number of Patients With Grade III-IV Acute Graft-versus-host Disease (aGVHD).
Description: Toxicity (undesireable effect) of this stem cell transplant preparative regimen due to acute graft-versus-host disease.
Time Frame: Day 100 Post Transplant
Measure: Number; unit: Participants
Arm/Group | Transplant Patients
Number analyzed (Participants) | 41
Participants | 2

ADVERSE EVENTS:
Arm/Group | Transplant Patients
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

LIMITATIONS AND CAVEATS:
Based on variability in age, diagnosis and condition of these patients, the data on enzyme levels and neuropsych testing is extremely difficult to report.

See Secondary Outcome Measures #3 and #4; no other adverse events were collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes